CLINICAL TRIAL: NCT02243761
Title: Canadian Institutes of Health Research (CIHR) Team in Innovations in Child and Youth Concurrent Disorders: Service Delivery and Treatment Subproject
Brief Title: Evaluating a Peer-Facilitated Skills-Based Intervention for Caregivers of Concurrent Disordered Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Childrens Centre Thunder Bay (Unknown)
Responsible Party: Principal Investigator, Shelley McMain, Head, Borderline Personality Disorder Clinic, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 129/2012
Record Dates: First submitted 2014-06-24; First posted 2014-09-18 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Caregiver Burden
Keywords: Concurrent Disorders; Mental Health; Addictions; Caregiver Burden
MeSH Terms: conditions — Caregiver Burden; Psychological Well-Being; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBT Based Skills Groups for Families (Experimental): Family members of youth with concurrent disorder participate in a 12-week DBT based skills group led by therapists and/or peer facilitators.
  Interventions: Other: DBT Based Skills Groups for Families

INTERVENTIONS:
Other: DBT Based Skills Groups for Families — 12 weeks of Dialectical Behaviour Therapy skills training group for families (90-minute once-weekly sessions)

SUMMARY:
Families of adolescents struggling with comorbid mental illness and addiction problems typically experience considerable emotional, financial and social burdens. Concurrent disorders (CDs) within families contribute to added stress and interpersonal conflict, as well as disrupt normal routines such as social and occupational activities. Despite the difficulties associated with being a family member of youth with CD, current mental health and addictions practices neglect to address this population. The overall purpose of this project is to assess the feasibility and clinical effectiveness of a Dialectical Behaviour Therapy skills (DBT) based training group for families of youth with CDs. The following main hypothesis will be examined: Family members of youth with concurrent disorders who participate in a 12-week skills group led by therapists and/or peer facilitators will show reduced caregiver burden and parenting stress from pre to post treatment.

DETAILED DESCRIPTION:
This study is designed to assess whether a 12-week skills based intervention is feasible and effective in addressing issues experienced by families of youth with concurrent mental health and addiction problems. Eligible subjects will be invited to participate in the following intervention:

The intervention is based on a DBT skills training model for families, the Family Connections© model. This model was originally developed for families of individuals with Borderline Personality Disorder (BPD) and later adapted for this study for CD.The Family Connections model is a 12-week (90-minute once-weekly sessions) skills training group designed to be led by therapists and/or peer support facilitators. The family groups in this study will be facilitated by two family members with experience being part of a family group and training and they will work with or without a professional therapist. Groups will consist of a maximum of 16 family members. Family members will receive a manual which describes the skills to be covered.

The skills-training will be delivered in two cities in collaboration with two organizations: CAMH, Toronto and the Children's Centre Thunder Bay. Participants will be recruited through advertisements posted on flyers and relevant websites.

The family intervention will evaluate change over time and use a mixed between/within subject, pre/post and follow-up design. Assessments will occur at baseline, mid-skills training (4 weeks), after 12-week skills training (post intervention), and at 12-week post intervention follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* literacy in English,
* are family members of an adolescent scoring in the clinical range on at least one subscale of the Child Behavior Checklist (CBCL)

Exclusion Criteria:

* has adolescent children participating in the sister youth intervention protocol #069-2011.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Family member burden & psychological stress as measured by the Burden Assessment Scale | Baseline, Mid-intervention (4 weeks post-baseline), Post-intervention (12 weeks post baseline), and at 12 weeks follow-up
  The primary outcome measure will examine change in family member burden and stress from baseline on standardized assessment instruments

CONTACTS AND LOCATIONS:
Overall Officials: Shelley McMain, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada